CLINICAL TRIAL: NCT07292909
Title: Randomized Trial to Evaluate the Anti-inflammatory Effects of Empagliflozin Following PCI
Brief Title: Effect of Empagliflozin on Inflammation
Acronym: EMPANTINFLAM
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hotel Dieu de France Hospital (Other)
Responsible Party: Principal Investigator, Rabih Azar, Professor of Medicine, Hotel Dieu de France Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEHDF 2511
Record Dates: First submitted 2025-12-06; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: CAD - Coronary Artery Disease; Inflamation; PCI; SGLT 2 Inhibitors
Keywords: CAD; inflammation; SGLT2 inhibitors
MeSH Terms: conditions — Coronary Artery Disease; Inflammation | interventions — empagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- empagliflozin (Active Comparator): Patients who will receive empagliflozin
  Interventions: Drug: Empagliflozin (SGLT2i)
- Placebo (Placebo Comparator): Placebo control
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Empagliflozin (SGLT2i) — Patient will receive 10 mg of empagliflozin PO per day, starting at least 2 days before planned PCI and on the day of PCI. Patient will thus receive at least 3 doses of empagliflozin prior to intervention
  Arms: empagliflozin
Drug: Placebo — Patient will receive a matching placebo PO 1 tab per day, starting at least 2 days before planned PCI and on the day of PCI. Patient will thus receive at least 3 doses of empagliflozin prior to intervention
  Arms: Placebo

SUMMARY:
Empagliflozin is a drug given to lower glucose. It is used in the treatment of diabetes. However, it was shown to improve symptoms and survival of patients who are suffering from heart failure. The exact mechanism of this effect is currently not clearly understood.

He hypothesize that empagliflozin has other properties than glucose lowering, that can explain its efficacy. One of these properties, is an anti-inflammatory effect.

To document this, we are using a model of inflammation following percutaneous coronary scenting. We know that patients who get a stent will develop inflammation following stenting. This is documenting by a higher level of C-Reactive Protein 24 hours after the procedure.

Patients who will participate in the study, will receive empagliflozin or a placebo tablet for 3 days prior to the revascularisation procedure. CRP and other inflammatory markers will be measured before intervention and 24 hours later. The goal is to demonstrate a lower rise in CRP following intervention in patients treated with empagliflozin vs. those who have received a placebo.

ELIGIBILITY:
Inclusion Criteria:

* • Patients with stable CAD who are electively scheduled for PCI on a de novo lesion in a native coronary artery

Exclusion Criteria:

* • Patients who have been taking an SGLT-2 inhibitor during the last month

  * Patients who are receiving any anti-inflammatory medication: immunosuppressor, steroids, NSAID…
  * Patients who have underlying inflammatory conditions such as rheumatic arthritis, infection, active malignancy
  * Patients with an acute coronary syndrome within the last month
  * Intervention on a restenotic lesion or lesion in a saphenous vein graft
  * Creatinine clearance less than 30 mL/min
  * Patients who are treated with devices other than balloons and stents (lithotripsy, rotational atherectomy…)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
CRP change | baseline and 18-24 hours after pci
  High sensitivity CRP will be measured immediately before and 18-24 hours after PCI

CONTACTS AND LOCATIONS:
Overall Officials: Rabih R Azar, MD, MPH, Principal Investigator — Hotel Dieu de Frace
Locations (1):
- Hotel Dieu de France, Beirut, Beyrouth, Lebanon

IPD SHARING:
Plan to Share IPD: Yes
We can share all patients data: demographics, characteristics of intervention, markers levels before and after the procedure
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: At end of study and for at least 3 years after completion
Access Criteria: Investigators, journal editors. They can contact us via email